CLINICAL TRIAL: NCT06773000
Title: Can Complex Carbohydrates and Essential Amino Acid Supplementation Improve Outcomes Following Geriatric Hip Fractures
Brief Title: Nutritional Supplementation in Geriatric Hip Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-00895
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Geriatric Hip Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XR™ Recovery Supplement (Experimental): 2 packets of XR Carbohydrate Loading will be administered the evening before surgery and one packet on the day of surgery up to 2 hours prior to the scheduled operating time. Participants will then take the XR™ Recovery Supplement twice daily for three weeks following their surgery.
  Interventions: Dietary Supplement: XR™ Recovery Supplement; Dietary Supplement: XR Carbohydrate Loading Supplement
- Standard nutritional counseling (No Intervention): The control group will receive standard of care nutritional counseling with a registered dietician once during inpatient admission, without the use of the supplement.

INTERVENTIONS:
Dietary Supplement: XR™ Recovery Supplement — Participants will receive a total daily dosage of 59.2 grams of XR™ Recovery Supplement orally, divided into two doses of 29.6 grams each (or two pouches). The dosing regimen will begin upon hospital admission and continue for three weeks post-operatively.
  Arms: XR™ Recovery Supplement
Dietary Supplement: XR Carbohydrate Loading Supplement — 2 packets of XR Carbohydrate Loading will be administered the evening before surgery and one packet on the day of surgery up to 2 hours prior to the scheduled operating time. The powder will be mixed with 14 oz of room temperature water only until dissolved then may be served over ice for desired temperature of consumption by the participant.
  Arms: XR™ Recovery Supplement

SUMMARY:
This study is a randomized controlled trial comparing outcomes between geriatric hip fractures who received a commercially available (XR RecoveryTM, Salt Lake City Utah) peri-operative nutritional supplement for three weeks post-operatively to those who receive standard nutritional counseling. The main question it aims to answer is:

- Does supplementation decrease muscle loss via ultrasound measurements of the cross-sectional area of the rectus femoris of the uninjured leg?

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 65 years or older.
2. Presenting with a geriatric hip fracture (femoral neck, intertrochanteric, or subtrochanteric) requiring surgical intervention.
3. Able to provide informed consent.
4. Expected to survive at least 6 months after surgery, with no terminal illness.

Exclusion Criteria:

1. Pre-existing conditions that significantly impair mobility prior to injury.
2. Severe renal or liver impairment.
3. Active treatment with investigational drugs or participation in another clinical trial within the last 30 days.
4. Inability to tolerate oral nutritional supplementation due to gastrointestinal disorders.
5. Allergies to any components of the nutritional supplement being tested.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change in muscle loss, as measured by the cross-sectional area of the rectus femoris muscle | Baseline, Visit 7 (1 year post operation)
  Outcome measure will be measured using ultrasound imaging.

SECONDARY OUTCOMES:
Number of inpatient complications related to the surgical procedure for hip fractures | From admission (visit 1) until discharge (~72 hours post-operation)
Number of wound complications | Visit 5, up to 6 months
  Complications include infection and bleeding.
Length of hospital stay | From admission (visit 1) until discharge (~72 hours post-operation)
Rate of readmission | Visit 7 (1 year post operation)
Mortality Rate | Visit 7 (1 year post operation)
Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) score | Baseline, Visit 7 (1 year post operation)
  A PROMIS PF score is a measurement of physical function that ranges from 0 to 100. The average score is 50, with a standard deviation of 10. A score of 40 is considered below average, indicating decreased physical function, while a score of 60 is considered above average, which indicates increased physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Ganta, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
REDCap data will be reshared with study sponsor in the form of de-identified aggregate data. Data collected for this study will be analyzed and stored at NYU Langone. After the study is completed, any identifiable information collected during the study will not be used or distributed for future research studies.